CLINICAL TRIAL: NCT03878394
Title: Comparison of the Effectiveness of Different Home Exercise Programs in Healthy Individuals
Brief Title: Comparison of the Effectiveness of Different Home Exercise Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10840098-604.01.01-E47630
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2019-03

CONDITIONS: Cognitive Function 1, Social
Keywords: balance; cognitive function; healthy individuals; quality of life; cognitive exercises; depression
MeSH Terms: conditions — Depression | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): The first group will be prescribed aerobic exercise and balance exercises as home exercise. Participants in this group will perform 30 min moderate walking exercises and balance exercises. Balance exercises shall consist of feet static stops for 30 second , one leg stance for 30 second, standing at tandem position for 30 second and uplift exercises at the fingertips for 30 second. Exercises will be held once a day for 3 days per week over 6 weeks.
  Interventions: Other: aerobic exercise and balance exercises
- Group 2 (Experimental): The second group will be prescribed cognitive tasks combined with aerobic exercise and balance exercises as home exercises. Participants in this group will have 30 minutes of moderate intensity exercise and cognitive tasks combined with balance exercises. Participants will be asked to count backwards from 20 during the walk and then count back the days of the week back and repeat it for 30 minutes. Balance exercises shall consist of feet static stops for 30 second , one leg stance for 30 second, standing at tandem position for 30 second and uplift exercises at the fingertips for 30 second. Patients will be asked to count backwards from 20 to count the days of the week backwards during balance exercises. Exercises will be held once a day for 3 days per week over six weeks. Participants will be called by the researcher on the days of the exercise and the participant's compliance with the exercise program will be checked.
  Interventions: Other: aerobic exercise and balance exercises; Other: aerobic exercise and balance exercises with cognitive exercises

INTERVENTIONS:
Other: aerobic exercise and balance exercises — The first group will be prescribed aerobic exercise and balance exercises as home exercise. Participants in this group will perform 30 min moderate walking exercises and balance exercises. Balance exercises shall consist of feet static stops for 30 second , one leg stance for 30 second, standing at tandem position for 30 second and uplift exercises at the fingertips for 30 second. Exercises will be held once a day for 3 days per week over 6 weeks.Exercise will be held once a day for 3 days per week over six weeks. Participants will be called by the researcher on the days of the exercise and the participant's compliance with the exercise program will be checked.
Other: aerobic exercise and balance exercises with cognitive exercises — The second group will be prescribed cognitive tasks combined with aerobic exercise and balance exercises as home exercises. Participants in this group will have 30 minutes of moderate intensity exercise and cognitive tasks combined with balance exercises. Participants will be asked to count backwards from 20 during the walk and then count back the days of the week back and repeat it for 30 minutes. Balance exercises shall consist of feet static stops for 30 second , one leg stance for 30 second, standing at tandem position for 30 second and uplift exercises at the fingertips for 30 second. Patients will be asked to count backwards from 20 to count the days of the week backwards during balance exercises. Exercises will be held once a day for 3 days per week over six weeks. Participants will be called by the researcher on the days of the exercise and the participant's compliance with the exercise program will be checked.
  Arms: Group 2

SUMMARY:
Aging is defined as a functional change in the organism which is not reversible with time progression. With this change in the organism, physical and cognitive functions are decreasing, and the potential of the individual to establish a balance between the systems decreased. For this reason, the aim of this is to investigate the effects of different home exercise programs on cognitive function, balance and daily living activities in healthy individuals.

DETAILED DESCRIPTION:
40 healthy individuals between the ages of 60-80 who agreed to participate in the study will be included in the study. Participants will be divided into 2 groups randomly. Both groups will be given balance exercises with aerobic exercise. The second group will be given second additional cognitive task besides doing usual exercises that the first group is performing. Exercises will be given in the form of a home exercise program and the treatment will last for 6 weeks. The continuity of the exercises will be controlled by telerehabilitation method. The participants will be evaluated before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 60 and 80
* Mini Mental Status Test score to be over 24

Exclusion Criteria:

* Cardiovascular disease
* Cardiovascular surgery operation, pacemaker etc.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MOCA) | 6 weeks
  Montreal Cognitive Assessment (MOCA) was developed by Nasreddine et al. to distinguish healthy individuals from individuals with mild cognitive impairment. MOCA evaluates 8 different functions including attention and concentration, executive functions, memory, language, visual-spatial skills, calculation and orientation and abstract thinking. The highest score is 30. 21 points and above are considered normal.
Stroop Test | 6 weeks
  The Stroop Test measures the speed of information processing, the ability to suppress a customary behavior, focused attention, the ability to perform an unusual behavior, and the ability to change perceptual setup under varying demands and under a disturbing effect. The standardization studies of Stroop Test in our country were performed by Karakaş et al. The Turkish form was named Stroop Test TBAG Form. The Stroop Test TBAG Form consists of four white cards. Each card has 6 rows sorted randomly and 4 items per line. These cards contain the stimulants of the test.
Benton Face Recognition Test | 6 weeks
  The face recognition test was developed by Benton in 1969. It is standardized to determine the capacity to identify and distinguish unrecognized human faces. This test consists of 22 pages of A4 size and there are face pictures on these pages. Only one page of pages is numbered. There is a stimulant picture on pages with no page numbers. Numbered pages have 6 pictures to select from among the responses. The application period of the test is 5-15 minutes and the time factor is not evaluated separately.

SECONDARY OUTCOMES:
Berg Balance Test | 6 weeks
  The reliability and validity of the Turkish form was performed by Şahin et al. The Berg Balance Test was designed to assess the balance in elderly adults and to determine the risk of falling. It is performed using a five-point scale to give scores to the subjects performing the fourteen functional activities. The maximum score in the Berg Balance Test is 56.A score below 40 indicates a reduction of approximately 100%.
6 Minute Walk Test | 6 weeks
  The 6 Minute Walk Test (6DYT) was adapted by American Thoracic Society (ATS) from the "12-Minute Cooper Test" developed by Cooper et al. It is used to evaluate the functional capacity of the person. This test measures the distance a patient can walk on a flat and hard surface for 6 minutes.
Geriatric Depression Scale | 6 weeks
  Geriatric Depression Scale was developed in 1983 by Yesavage et al. Turkish validity and reliability study was conducted in 1997 by Ertan et al. Geriatric Depression Scale consists of 30 questions based on self-report and questions are answered yes or no. Each response with a symptom of depression is evaluated as one point.
Short Form 36 Quality of Life Questionnaire (SF-36) | 6 weeks
  The SF-36 is a general health screening survey designed in America. The reliability and validity of the SF-36 were performed by Koçyiğit et al. in 50 patients with osteoarthritis and 50 patients with low back pain. Questions examine 8 different subgroups of health. It also includes the physical activity limitations perceived by the patient.
Time up and Go Test | 6 weeks
  Time up and Go Test was developed in 1991 by Diane et al. This test evaluates the risk of falling and mobility in the elderly. Time up and Go Test is a balance and gait index that requires the patient to stand up from a chair, walk 3 meters, return to the chair and sit down. The time required to complete the task is measured in seconds.
Mini Mental Durum Test | 6 weeks
  The Mini Mental Test (MMT) was developed in 1975 by Folstein. It consists of 11 questions evaluating cognitive functions such as test, recall, language, record memory, calculation, orientation. The applicability and reliability of this test has been enhanced by the Standardized Practice Guide developed by Molloy et al. The MMT is divided into two parts, the first part only requires a voice response and includes orientation, memory and attention; the highest score is 21. The second section tests name capability, follow verbal and written commands and single-handedly write the sentence . It involves copying a complex polygon similar to the Bender-Gestalt Figure. The maximum score is 9.

CONTACTS AND LOCATIONS:
Overall Officials: Miray Budak, assoc.prof., Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Beykoz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu-Ambrose T, Nagamatsu LS, Graf P, Beattie BL, Ashe MC, Handy TC. Resistance training and executive functions: a 12-month randomized controlled trial. Arch Intern Med. 2010 Jan 25;170(2):170-8. doi: 10.1001/archinternmed.2009.494. PMID 20101012
- [Background] Nagamatsu LS, Handy TC, Hsu CL, Voss M, Liu-Ambrose T. Resistance training promotes cognitive and functional brain plasticity in seniors with probable mild cognitive impairment. Arch Intern Med. 2012 Apr 23;172(8):666-8. doi: 10.1001/archinternmed.2012.379. No abstract available. PMID 22529236
- [Background] Paterson DH, Warburton DE. Physical activity and functional limitations in older adults: a systematic review related to Canada's Physical Activity Guidelines. Int J Behav Nutr Phys Act. 2010 May 11;7:38. doi: 10.1186/1479-5868-7-38. PMID 20459782
- See also: Pubmed Link — https://www.ncbi.nlm.nih.gov/pubmed/20101012
- See also: Pubmed Link — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3514552/
- See also: Pubmed Link — https://www.ncbi.nlm.nih.gov/pubmed/20459782